CLINICAL TRIAL: NCT06744465
Title: NearWave Optical Molecular Monitoring for Predicting Complete Pathological Response (pCR) to Neoadjuvant Chemotherapy (NAC) in Breast Cancer Patients
Brief Title: NearWave Optical Molecular Monitoring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: University of Notre Dame (Other); Elevate Ventures (Unknown); NearWave Corp. (Unknown)
Responsible Party: Principal Investigator, Tarah J Ballinger, MD, Assistant Professor of Clinical Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CTO-IUSCCC-0880
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer; TNBC - Triple-Negative Breast Cancer; HER2-negative Breast Cancer; Invasive Breast Carcinoma
Keywords: neoadjuvant chemotherapy; breast cancer; imaging; NearWave; invasive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- NearWave monitoring (Experimental): Breast cancer patients receiving neoadjuvant chemotherapy treatment followed by surgery will be monitored by a noninvasive handheld imaging device before, during and after chemotherapy.
  Interventions: Device: NearWave monitoring

INTERVENTIONS:
Device: NearWave monitoring — NearWave optical molecular monitoring

SUMMARY:
The purpose of this study is to assess the feasibility of the NearWave optical molecular monitoring system for monitoring therapy progression and predicting pathologic complete response (pCR) of breast cancer patients undergoing neoadjuvant chemotherapy (NAC).

DETAILED DESCRIPTION:
This is a prospective, observational, pilot study. Due to the investigational nature of the NearWave device, imaging data collected will not be used to inform patient treatment. Since this is our first experience with the NearWave device and there does not exist any preliminary data with this device, we are performing this pilot study to establish whether data collected is of high enough quality to warrant further study.

Primary Objective: The primary objective of this study is to assess the feasibility of using the NearWave optical molecular monitoring system during therapy to predict pCR in breast cancer patients undergoing NAC, measured by the data quality captured with the device.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Patients who:

   1. have been diagnosed with invasive breast cancer by tissue biopsy and have not yet started any therapy for the disease; a) Subtype HER2 positive (IHC 3+ or if IHC 2+, then positive by FISH), with any ER status, OR b) Subtype TNBC, defined by: HER2 negative and ER/PR negative or low (ER and PR ≤ 9%, weak staining)
   2. with ≥2 cm tumor size in the largest dimension as measured by ultrasound, MRI, or mammography. If multifocal disease, at least one tumor must measure ≥2 cm
   3. are planned to receive neoadjuvant chemotherapy followed by surgery
   4. Will be at least two weeks out from biopsy of the primary lesion at the time of baseline visit
   5. Have a palpable breast mass as determined by a treating physician

Exclusion Criteria:

1. Patients with significant bruising or hematoma from diagnostic breast biopsy, as determined by clinical judgement (mild ecchymosis okay)
2. Inflammatory breast cancer
3. Prior breast cancer requiring surgery or radiation in either breast
4. Pregnant or nursing due to changes in breast architecture
5. Patients with a BMI of ≥ 40, unless the lesion is near the surface (<3 cm from the skin surface), based on diagnostic scan measurements
6. Patients with any tattoos on their breasts

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using NearWave imaging as a monitoring system | Over approximately 5 months; baseline, mid way through treatment, and at last dose of clinical chemotherapy/prior to clinical surgery
  Adequate data quality metrics:
  Signal-to-noise ratio (SNR) (measurement that compares the strength of a signal to the level of background noise) above 10 dB for at least 80% of collected data points;
Feasibility of using NearWave imaging as a monitoring system | Over approximately 5 months; baseline, mid way through treatment, and at last dose of clinical chemotherapy/prior to clinical surgery
  Adequate data quality metrics:
  • Model fit metric: Root mean squared error (RMSE) ( the average difference between the predicted values and the actual values) of 5x10-4 or lower for regressions of calibrated imaging
Feasibility of using NearWave imaging as a monitoring system | Over approximately 5 months; baseline, mid way through treatment, and at last dose of clinical chemotherapy/prior to clinical surgery
  Adequate data quality metrics:
  • Estimated tissue concentrations of HHb, HbO2, water, and lipid within expected physiological ranges.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided